CLINICAL TRIAL: NCT06508281
Title: Investigation of the Effect of Model Video Activity on Medical Faculty Students' Anatomy Education
Brief Title: Model Video Activity in Anatomy Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Giresun University (Other)
Responsible Party: Principal Investigator, NAkbayturk, PhD, Assistant Professor, Giresun University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: GRU-ANA-NA-01
Record Dates: First submitted 2024-07-09; First posted 2024-07-18 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Anatomy; Medical Students; Education
Keywords: anatomy; education; medical students; learning

STUDY DESIGN:
Intervention Model Description: it was planned to conduct a randomized controlled trial on the effect of model video activity in anatomy education on the anatomy education of medical faculty students in a pretest-posttest order.
Who Masked: Participant
Masking Description: Students who agreed to participate in the study were divided into experimental and control groups using the randomization method.
  It consisted of 148 students studying in the first grade. There were students who did not meet the study criteria and did not take the pre-tests and post-tests. As a result, 95 participants were included in the study, 46 in the experimental group and 49 in the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): After the anatomy course topic is explained in class, students will answer the theoretical questions about the subjects and the pre-test online via a Google Forms survey. Anatomy model videos prepared by the researchers for the experimental group students will be uploaded to Google Drive and sent via link. Students will be asked to log in from their computer or mobile phone and watch anatomy model videos whenever and wherever they want. Students in the experimental group will answer the final test after studying for a week and watching videos on Facial Muscles, Neck Anatomy and Muscles (Anterior Side Region Muscles and Triangles), Forearm Anterior Region Muscles, Forearm Posterior Region Muscles and Hand Muscles.
  Interventions: Other: experimental group
- control group (No Intervention): No application will be made to the control group and their training will continue only with the traditional method. Control group students will fill out the theoretical questions test again on the topics "Facial Muscles, Neck Anatomy and Muscles (Anterior Side Region Muscles and Triangles), Forearm Anterior Region Muscles, Forearm Posterior Region Muscles and Hand Muscles

INTERVENTIONS:
Other: experimental group — . Anatomy model videos prepared by the researchers for the experimental group students will be uploaded to Google Drive and sent via link. Students will be asked to log in from their computer or mobile phone and watch anatomy model videos whenever and wherever they want
  Arms: experimental group

SUMMARY:
During Anatomy education and training at medical school; In addition to theoretical lecture presentations, visual alternative methods such as videos can be used to better understand, learn and keep in mind anatomical structures, to help reinforce knowledge and to increase students' motivation in anatomy lessons. Model videos can be an alternative to visual anatomy education in order to provide a better understanding of the subjects so that people can watch model videos wherever and whenever they want, in addition to the theoretical lesson.

DETAILED DESCRIPTION:
The study aims to evaluate the effect of using model video activity on anatomy education in first-year medical faculty students. This study was planned to be conducted in a randomized controlled trial in a pre-test-post-test design to determine the effect of model video activity in anatomy education on the anatomy education of medical faculty students.The population of the research will be first-year students at Giresun University Faculty of Medicine, and the sample will be students who agree to participate in the research. Students who agreed to participate in the study were divided into experimental and control groups using the randomization method. Participants' consent to participate in the study was obtained by ticking the 'Volunteer consent form' and 'I want to participate in the study' box on the first page of the survey. Students who accept the research will fill out the "Introductory Characteristics of Students Form". After the anatomy course topic is explained in class, students will answer the theoretical questions about the subjects and the pre-test online via a Google Forms survey. Anatomy model videos prepared by the researchers for the experimental group students will be uploaded to Google Drive and sent via link. Students will be asked to log in from their computer or mobile phone and watch anatomy model videos whenever and wherever they want. Students in the experimental group will answer the final test after studying for a week and watching videos on Facial Muscles, Neck Anatomy and Muscles (Anterior Side Region Muscles and Triangles), Forearm Anterior Region Muscles, Forearm Posterior Region Muscles and Hand Muscles.

No application will be made to the control group and their training will continue only with the traditional method. Control group students will fill out the theoretical questions test again on the topics "Facial Muscles, Neck Anatomy and Muscles (Anterior Side Region Muscles and Triangles), Forearm Anterior Region Muscles, Forearm Posterior Region Muscles and Hand Muscles".

After the experimental group application is completed and all data is received, anatomy model videos will be shared with the control group students. Students will be asked to fill out the 'Anatomy Model Video Activity Feedback Form'.

ELIGIBILITY:
Inclusion Criteria:

* First year students of Giresun University Faculty of Medicine
* Students who volunteered to participate in the study

Exclusion Criteria:

* Giresun University Faculty of Medicine 2nd, 3rd, 4th, 5th and 6th grade students
* Students who do not have a smartphone or computer and do not have internet access
* Students who did not volunteer to participate in the study

Ages: 17 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 148 (Actual)
Dates: Start 2024-04-04 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2024-05-25 (Actual)

PRIMARY OUTCOMES:
The effects of model video activity in anatomy education on the anatomy education of medical faculty students were measured with the 'Anatomy theoretical questions test' prepared by the researchers. | The duration of watching anatomy model videos for each subject is 1 week. The time to complete the 'Anatomy theoretical questions test' pre-tests and post-tests is 1 week each.
  A randomized controlled study with pre-test-post-test design with experimental and control groups. 'Anatomy theoretical questions test' prepared for pre-test and post-test was given to students before and after watching anatomy model videos. 'Anatomy theoretical questions test' prepared by researchers consists of 25 questions, each with five options.

CONTACTS AND LOCATIONS:
Locations (1):
- Giresun University, Faculty of Medicine, Department of Anatomy, Giresun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No